CLINICAL TRIAL: NCT00030719
Title: High Risk Neuroblastoma Study 1 Of Siop-Europe
Brief Title: Combination Chemotherapy With or Without Filgrastim Before Surgery, High-Dose Chemotherapy, and Radiation Therapy Followed by Isotretinoin With or Without Monoclonal Antibody in Treating Patients With Neuroblastoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069191; SIOP-EUROPE-HR-NBL-1; ESIOP; EU-20148
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2010-08

CONDITIONS: Neuroblastoma
Keywords: regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; dinutuximab; Busulfan; Carboplatin; Cyclophosphamide; Etoposide; Isotretinoin; Melphalan; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: monoclonal antibody Ch14.18
Drug: busulfan
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: isotretinoin
Drug: melphalan
Drug: vincristine sulfate
Procedure: bone marrow ablation with stem cell support
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. Combining chemotherapy with peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining isotretinoin and monoclonal antibodies may kill any remaining tumor cells following surgery. It is not yet known which treatment regimen is more effective in treating neuroblastoma.

PURPOSE: This randomized phase III trial is studying how well combination chemotherapy with or without filgrastim before surgery, high-dose chemotherapy, and radiation therapy followed by isotretinoin with or without monoclonal antibody work in treating patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of myeloablative therapy with busulfan and melphalan vs carboplatin, etoposide, and melphalan, in terms of 3- and 5-year event-free survival (EFS), progression-free survival (PFS), and overall survival (OS), in patients with high-risk neuroblastoma.
* Compare the 3-year EFS in these patients treated with isotretinoin with or without monoclonal antibody Ch14.18 after myeloablative therapy.
* Determine the response at metastatic sites after induction chemotherapy in these patients.
* Determine the effect of metastatic disease response after induction chemotherapy on EFS, PFS, and OS in these patients.
* Compare the toxicity and episodes of febrile neutropenia in patients treated with induction chemotherapy with or without filgrastim (G-CSF).
* Determine the effect of elective hematopoietic support with G-CSF during induction chemotherapy on peripheral blood stem cell collection in these patients.
* Compare the acute and long-term toxic effects of the 2 myeloablative therapy regimens in these patients.
* Determine the effect of radiotherapy on pre-surgical tumor volume at the primary site on local control, EFS, PFS, and OS in these patients.
* Determine the tolerability of isotretinoin with or without monoclonal antibody Ch14.18 after myeloablative therapy in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (2 or 3 with MycN amplification vs 4). Patients are randomized to 1 of 8 treatment arms:

Arm I:

* Patients receive induction chemotherapy comprising vincristine IV, carboplatin IV over 1 hour, and etoposide IV over 4 hours on days 1 and 41; vincristine IV and cisplatin IV over 24 hours on days 11, 31, 51, and 71; and vincristine IV on days 21 and 61 and cyclophosphamide IV and etoposide over 4 hours on days 21, 22, 61, and 62. Patients receive filgrastim (G-CSF) subcutaneously on days 3-8, 12-18, 23-28, 32-38, 43-48, 52-58, 63-68, and 72 until peripheral blood stem cell (PBSC) collection.
* Patients undergo PBSC collection beginning on day 80. Patients then undergo surgery on day 95.
* Patients receive myeloablative therapy comprising oral busulfan 4 times daily on days -6 to -3 and melphalan IV over 15 minutes on day -2. Patients undergo PBSC infusion on day 0.
* Patients undergo radiotherapy in 14 fractions over 21 days.
* Beginning within 30 days after radiotherapy, patients receive oral isotretinoin twice daily on days 1-14. Treatment repeats every 28 days for 6 courses.

Arm II:

* Patients receive induction chemotherapy as in arm I, but with no G-CSF. Patients then undergo PBSC collection and surgery as in arm I. Patients receive myeloablative therapy and undergo PBSC infusion as in arm I. Patients undergo radiotherapy as in arm I.
* Patients receive oral isotretinoin twice daily on days 1-14 and monoclonal antibody Ch14.18 IV over 8 hours on days 1-5. Treatment repeats every 28 days for 6 courses for isotretinoin and every 28 days for 5 courses for monoclonal antibody Ch14.18.

Arm III:

* Patients receive induction chemotherapy and G-CSF as in arm I. Patients then undergo PBSC collection and surgery as in arm I. Patients receive myeloablative therapy and undergo PBSC infusion as in arm I. Patients undergo radiotherapy as in arm I. Patients receive isotretinoin as in arm I.

Arm IV:

* Patients receive induction chemotherapy as in arm II. Patients then undergo PBSC collection and surgery as in arm I. Patients receive myeloablative therapy and undergo PBSC infusion as in arm I. Patients undergo radiotherapy as in arm I. Patients receive isotretinoin and monoclonal antibody Ch14.18 as in arm II.

Arm V:

* Patients receive induction chemotherapy and G-CSF as in arm I.
* Patients receive myeloablative therapy comprising carboplatin IV continuously and etoposide IV continuously on days -7 to -4 and melphalan IV over 15 minutes on days -7 to -5. Patients undergo PBSC infusion on day 0.
* Patients undergo radiotherapy as in arm I. Patients receive isotretinoin as in arm I.

Arm VI:

* Patients receive induction chemotherapy as in arm II. Patients receive myeloablative therapy and undergo PBSC infusion as in arm V. Patients undergo radiotherapy as in arm I. Patients receive isotretinoin and monoclonal antibody Ch14.18 as in arm II.

Arm VII:

* Patients receive induction chemotherapy and G-CSF as in arm I. Patients receive myeloablative therapy and undergo PBSC infusion as in arm V. Patients undergo radiotherapy as in arm I. Patients receive isotretinoin as in arm I.

Arm VIII:

* Patients receive induction chemotherapy as in arm II. Patients receive myeloablative therapy and undergo PBSC infusion as in arm V. Patients undergo radiotherapy as in arm I. Patients receive isotretinoin and monoclonal antibody Ch14.18 as in arm II.

Patients on all treatment arms are followed every 6 months for 3 years and then annually for 2 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: Approximately 175 patients per year will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma according to International Neuroblastoma Staging System

  * Stage 2 or 3 with MycN amplification
  * Stage 4
* Tumor material available for determination of biological prognostic factors

PATIENT CHARACTERISTICS:

Age:

* 1 to 20 at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 3 times normal
* ALT less than 3 times normal

Renal:

* Creatinine less than 1.5 mg/mL
* Creatinine clearance and/or glomerular filtration rate at least 60 mL/min

Cardiovascular:

* Shortening fraction at least 28% OR
* Ejection fraction at least 55%
* No clinical congestive heart failure

Pulmonary:

* Chest x-ray normal
* Oxygen saturation normal

Other:

* HIV negative
* No Brock grade 2 or greater
* No uncontrolled infections requiring IV antivirals, antibiotics, or antifungals
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 1 prior chemotherapy regimen for localized unresectable disease
* No concurrent anthracyclines
* No other concurrent chemotherapy

Endocrine:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent investigational therapy

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 175 (Estimated)
Dates: Start 2001-12

PRIMARY OUTCOMES:
Event-free survival at 3 years
Mean number of febrile events during induction

SECONDARY OUTCOMES:
Response rate assessed by the International Neuroblastoma Response Criteria after 4 and 8 induction chemotherapy courses
Event-free survival at 5 years
Overall survival
Toxicity
Biological factors (i.e., MycNM amplification, 1p deletion, ploidy, 17 q+, CD44, and Trk-A)
Serum concentrations of lactic dehydrogenase, ferritin, neurone specific enolase
Urinary catecholamines at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Ladenstein, MD, Study Chair — St. Anna Kinderkrebsforschung
Locations (32):
- St. Anna Children's Hospital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Aarhus Universitetshospital - Aarhus Sygehus, Aarhus, Denmark
- Institut Gustave Roussy, Villejuif, France
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Fondazione Istituto Nazionale dei Tumori, Milan, Italy
- Rikshospitalet University Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, SA, Lisbon, Portugal
- Hospital Universitario La Fe, Valencia, Spain
- Karolinska University Hospital - Solna, Stockholm, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Result] Ladenstein R, Valteau-Couanet D, Brock P, Yaniv I, Castel V, Laureys G, Malis J, Papadakis V, Lacerda A, Ruud E, Kogner P, Garami M, Balwierz W, Schroeder H, Beck-Popovic M, Schreier G, Machin D, Potschger U, Pearson A. Randomized Trial of prophylactic granulocyte colony-stimulating factor during rapid COJEC induction in pediatric patients with high-risk neuroblastoma: the European HR-NBL1/SIOPEN study. J Clin Oncol. 2010 Jul 20;28(21):3516-24. doi: 10.1200/JCO.2009.27.3524. Epub 2010 Jun 21. PMID 20567002
- [Derived] Veal GJ, Nguyen L, Paci A, Riggi M, Amiel M, Valteau-Couanet D, Brock P, Ladenstein R, Vassal G. Busulfan pharmacokinetics following intravenous and oral dosing regimens in children receiving high-dose myeloablative chemotherapy for high-risk neuroblastoma as part of the HR-NBL-1/SIOPEN trial. Eur J Cancer. 2012 Nov;48(16):3063-72. doi: 10.1016/j.ejca.2012.05.020. Epub 2012 Jun 26. PMID 22742881